CLINICAL TRIAL: NCT06437067
Title: A Real-world Study on the Long-term Prognosis of Acute-on-chronic Liver Failure
Brief Title: Study on Prognosis of Acute-on-chronic Liver Failure Complicated by Bacterial or Fungal Infection
Status: Recruiting | Type: Observational
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: ACLF-I
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-infection group: patients without bacterial or fungal infection
- bacterial infection group: patients with bacterial infection
- fungal infection group: patients with fungal infection

SUMMARY:
The subjects of this study were inpatients with ACLF who were admitted to Tongji Hospital in Wuhan from March 2023 to June 2025. After patients were enrolled, The patient's general information (gender, age, past medical history, etc.), complications (ascites, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding, etc.), laboratory tests (CRP, PCT, INR, WBC, fungal/bacterial diagnostic tests, etc.), symptoms and signs at the time of infection, and at admission (D1), D4, D7, D14, D21, etc.) were recorded Save the blood separately. The patients were divided into fungal infection group, bacterial infection group and non-infection group according to the infection status after admission.

ELIGIBILITY:
Inclusion Criteria:

1. TBIL ≥ 12 mg/mL and INR ≥ 1.5
2. Chronic hepatitis B

Exclusion Criteria:

(1) <18 or >80 years old; (2) primary hepatic or extrahepatic carcinoma; (3) with severe diseases of other organs or systems; (4) pregnancy; (5) imcomplete information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with ACLF admitted to Tongji Hospital in Wuhan from March 2023 to June 2025.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence rate of bacterial or fungal infection | 28 days and 90 days
  incidence rate of bacterial or fungal infection
mortality rate of bacterial or fungal infection | 28 days and 90 days
  mortality rate of bacterial or fungal infection

SECONDARY OUTCOMES:
incidence rate of complications | 28 days and 90 days
  incidence rate of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Disease, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China